CLINICAL TRIAL: NCT02503540
Title: Peripheral and Macular Retinal Vascular Perfusion and Leakage Dynamics in Diabetic Macular Edema and Retinal Venous Occlusions During Intravitreal Aflibercept Injection (IAI) Treatment for Retinal Edema: PERMEATE Study
Brief Title: Peripheral and Macular Retinal Vascular Perfusion and Leakage in DME and RVO
Acronym: PERMEATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Justis Ehlers (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Justis Ehlers, Assistant Professor of Ophthalmology, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-442
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Retinal Vein Occlusion; Diabetic Macular Edema; Branch Retinal Vein Occlusion; Central Retinal Vein Occlusion
Keywords: macular edema; rvo; diabetic macular edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Other): Monthly aflibercept for 6 months and then every other month for 6 months.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal aflibercept will be given q4 wks for 6 treatments and then q 8 weeks through month 12.
  Other Names: Eylea

SUMMARY:
This interventional study will evaluate the retinal vascular dynamics associated with Intravitreal Aflibercept Injection (IAI) therapy in eyes with diabetic macular edema (DME) or macular edema secondary to retinal vein occlusion (RVO). Ultra-widefield fluorescein angiography and optical coherence tomography (OCT) angiography will be performed at multiple timepoints to assess the changes in retinal vascular leakage, ischemia, and vascular abnormalities throughout the study duration and compare these alterations to baseline.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) and macular edema secondary to retinal venous occlusive diseases are the most common cause of vision loss from a retinal vascular disease. Recently, vascular endothelial growth factor (VEGF) inhibitors (bevacizumab, aflibercept, and ranibizumab) have been described as new first-line therapies for these conditions. Aflibercept is the most recently approved VEGF inhibitor for the management of these conditions. Clinical trials have shown that treatment with aflibercept improves visual acuity and reduces macular edema in a large percentage of patients.

This study will examine the changes that occur with intravitreal aflibercept to perfusion and leakage in treatment naive eyes over the course of 1 year.

ELIGIBILITY:
Inclusion Criteria

A subject must meet the following criteria to be eligible for inclusion in the study:

1. Signed Informed Consent.
2. Men and women ≥ 18 years of age.
3. Foveal-involving retinal edema secondary to DME or RVO based on investigator review of SDOCT.
4. E-ETDRS best-corrected visual acuity of: 20/25 to 20/400 in the study eye or Hand Motion (HM) in the study eye.
5. Willing, committed, and able to return for all clinic visits and complete all study related procedures.
6. Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) understand and willing to sign the informed consent form.

Exclusion Criteria

A subject who meets any of the following criteria will be excluded from the study:

1. Any prior or concomitant therapy with another investigational agent to treat DME or RVO in the study eye.
2. Prior panretinal photocoagulation in the study eye.
3. Prior intravitreal anti-VEGF therapy in the study eye.
4. Prior focal/grid laser photocoagulation in the study eye.
5. Prior history of intravitreal steroid therapy in the study eye.
6. Any history of allergy to fluorescein sodium or other reason that the patient is unable to undergo fluorescein angiography (e.g., inability to get vascular access, unable to tolerate procedure)
7. Prior systemic anti-VEGF therapy, investigational or FDA-approved, is only allowed up to 3 months prior to first dose, and will not be allowed during the study.
8. Significant vitreous hemorrhage obscuring view to the macula or the retinal periphery as determined by the investigator on clinical exam and ultra-widefield angiography.
9. Presence of other causes of macular edema, including myopic degeneration, ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, choroidal neovascularization, neovascular age-related macular degeneration or multifocal choroiditis in the study eye. Epiretinal membranes are allowed.
10. Presence of macula-threatening traction retinal detachment.
11. Prior vitrectomy in the study eye.
12. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
13. Any history of macular hole of stage 2 and above in the study eye.
14. Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as it's unlikely to interfere with the injection.
15. Prior trabeculectomy or other filtration surgery in the study eye.
16. Uncontrolled glaucoma at baseline evaluation (defined as intraocular pressure ≥25 mmHg despite treatment with anti-glaucoma medication) in the study eye.
17. Active intraocular inflammation in either eye.
18. Active ocular or periocular infection in either eye.
19. Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
20. Any history of uveitis in either eye.
21. Active scleritis or episcleritis in either eye.
22. Presence or history of scleromalacia in either eye.
23. Aphakia in the study eye.
24. Previous therapeutic radiation in the region of the study eye.
25. History of full-thickness penetrating keratoplasty in the study eye. Partial thickness corneal transplants including Descemet stripping automated endothelial keratoplasty and Descemet membrane endothelial keratoplasty are allowed.
26. Significant media opacities, including cataract, in the study eye which might interfere with visual acuity, assessment of safety, or fundus photography.
27. Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 52 week study period.
28. Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
29. Participation as a subject in any clinical study within the 12 weeks prior to Day 1.
30. Any systemic therapy with an investigational agent in the past 3 months prior to Day 1.
31. Any history of allergy to povidone iodine.
32. Pregnant or breast-feeding women
33. Women of childbearing potential* who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

    * Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justis P Ehlers, MD, Principal Investigator — Cole Eye Institute, Cleveland Clinic, OH 44195
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wessel MM, Nair N, Aaker GD, Ehrlich JR, D'Amico DJ, Kiss S. Peripheral retinal ischaemia, as evaluated by ultra-widefield fluorescein angiography, is associated with diabetic macular oedema. Br J Ophthalmol. 2012 May;96(5):694-8. doi: 10.1136/bjophthalmol-2011-300774. Epub 2012 Mar 15. PMID 22423055
- [Background] Thickett DR, Armstrong L, Millar AB. Vascular endothelial growth factor (VEGF) in inflammatory and malignant pleural effusions. Thorax. 1999 Aug;54(8):707-10. doi: 10.1136/thx.54.8.707. PMID 10413724
- [Background] Singer M, Tan CS, Bell D, Sadda SR. Area of peripheral retinal nonperfusion and treatment response in branch and central retinal vein occlusion. Retina. 2014 Sep;34(9):1736-42. doi: 10.1097/IAE.0000000000000148. PMID 24732695
- [Background] Rakic JM, Lambert V, Devy L, Luttun A, Carmeliet P, Claes C, Nguyen L, Foidart JM, Noel A, Munaut C. Placental growth factor, a member of the VEGF family, contributes to the development of choroidal neovascularization. Invest Ophthalmol Vis Sci. 2003 Jul;44(7):3186-93. doi: 10.1167/iovs.02-1092. PMID 12824270
- [Background] Ferrara N. Vascular endothelial growth factor and the regulation of angiogenesis. Recent Prog Horm Res. 2000;55:15-35; discussion 35-6. PMID 11036931
- [Background] Ferrara N, Houck KA, Jakeman LB, Winer J, Leung DW. The vascular endothelial growth factor family of polypeptides. J Cell Biochem. 1991 Nov;47(3):211-8. doi: 10.1002/jcb.240470305. PMID 1791185
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Derived] Figueiredo N, Srivastava SK, Singh RP, Babiuch A, Sharma S, Rachitskaya A, Talcott K, Reese J, Hu M, Ehlers JP. Longitudinal Panretinal Leakage and Ischemic Indices in Retinal Vascular Disease after Aflibercept Therapy: The PERMEATE Study. Ophthalmol Retina. 2020 Feb;4(2):154-163. doi: 10.1016/j.oret.2019.09.001. Epub 2019 Sep 10. PMID 31757691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from within ophthalmology clinics.
Pre-assignment Details: Single arm study.
Period: Overall Study
Arm/Group | Aflibercept
Started | 31
Completed | 28
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
Arm/Group | Aflibercept
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  years
    number analyzed (Participants) | 29
    (all) | 67.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  Participants
    number analyzed (Participants) | 29
    Female | 11
    Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  Participants
    number analyzed (Participants) | 29
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 6
    White | 23
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Measure Analysis Population Description: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  participants
    United States: number analyzed (Participants) | 29
    United States | 29
Baseline best corrected visual acuity [Mean (Standard Deviation); unit: ETDRS letters] — Population: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  ETDRS letters
    number analyzed (Participants) | 29
    (all) | 54.3 (23.3)
Baseline central subfield thickness [Mean (Standard Deviation); unit: μm] — Population: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  μm
    number analyzed (Participants) | 29
    (all) | 541.2 (242.3)
Panretinal leakage index [Mean (Standard Deviation); unit: percent] — Percentage of area of the visible retina that was leaking Population: Measure Analysis Population Description: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  percent
    number analyzed (Participants) | 29
    (all) | 3.4 (3.8)
Panretinal ischemic index [Mean (Standard Deviation); unit: percent] — Population: Measure Analysis Population Description: The PERMEATE study included 31 eyes. Two participants did not continue the study past month 3 because of elective study withdrawal (n = 1) and death (n = 1). Thus, 29 participants were included in the analysis.
  percent
    number analyzed (Participants) | 29
    (all) | 5.5 (8)
Number of patient with visual acuity of 20/200 or worse [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Panretinal Leakage Index at Month 12 From Baseline
Description: Change in panretinal leakage index (defined as the proportion of retinal area involved in angiographic leakage) at month 12 from baseline as measured by ultra-widefield angiography (UWFA).
Time Frame: 12 months
Population: Monthly aflibercept for 6 months and then every other month for 6 months.
Measure: Mean (Standard Deviation); unit: percentage of region of interest in UWFA
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
percentage of region of interest in UWFA | -3.14 (0.03)

2. Secondary Outcome: Mean Change in Total Leakage Index
Description: Mean change in total leakage index from baseline to month 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of region of interest in UWFA
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
percentage of region of interest in UWFA | 0.47 (2.0)

3. Secondary Outcome: Change in Panretinal Ischemic Index
Description: Change in panretinal ischemic index from baseline to postoperative month 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of region of interest in UWFA
Arm/Group | Aflibercept
Number analyzed (Participants) | 28
percentage of region of interest in UWFA | 3.2 (0.12)

4. Secondary Outcome: Change in Panretinal Ischemic Index From Baseline at 6 Months
Description: Change in panretinal ischemic index (defined as the proportion of retinal area with nonperfusion) from baseline at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of region of interest in UWFA
Arm/Group | Aflibercept
Number analyzed (Participants) | 28
percentage of region of interest in UWFA | 0.67 (0.03)

5. Secondary Outcome: Mean Change From Baseline Central Subfield Thickness
Description: OCT central subfield thickness change from baseline to 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
μm | 278.0 (251.3)

6. Secondary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA) Score Based on ETDRS
Description: Mean change from baseline in best-corrected visual acuity (BCVA) score from baseline to month 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
ETDRS letters | 18.4 (21.4)

7. Secondary Outcome: Number of Participants Who Gained 15 ETDRS Letters or More of Vision
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 13

8. Secondary Outcome: Number of Patients Who Gained 15 ETDRS Letters or More of Vision
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 12

9. Secondary Outcome: Number of Patients That Showed Visual Acuity 20/40 or Better
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 20

10. Secondary Outcome: Number of Patients That Showed Visual Acuity 20/200 or Worse
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 2

11. Secondary Outcome: Ocular Serious Adverse Events
Time Frame: 12 months
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 31
Participants | 0

12. Secondary Outcome: Number of Participants Who Lost 15 ETDRS Letters or More of Vision
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 1

13. Secondary Outcome: Number of Participants Who Lost 15 ETDRS Letters or More of Vision
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 0

14. Secondary Outcome: Number of Patients That Showed Visual Acuity 20/40 or Better
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 19

15. Secondary Outcome: Number of Patients That Showed Visual Acuity 20/200 or Worse
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
Participants | 0

16. Secondary Outcome: Mean Change From Baseline Central Subfield Thickness
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Aflibercept
Number analyzed (Participants) | 29
μm | 301.3 (250.3)

17. Secondary Outcome: Systemic Serious Adverse Events
Description: Incidence of systemic SAEs
Time Frame: 12 Months
Population: All subjects enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 31
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aflibercept
All-Cause Mortality (participants affected / at risk) | 2/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept (N=31)
Death (General disorders) | 2
Stroke (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT02503540/Prot_SAP_000.pdf